CLINICAL TRIAL: NCT06189313
Title: A Prospective, Multicenter Study to Evaluate the Safety and Efficacy of an Aspiration Thrombectomy System in Acute Pulmonary Embolism
Brief Title: CLEANer Aspiration for Pulmonary Embolism
Acronym: CLEAN-PE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Argon Medical Devices (Industry)
Collaborators: NAMSA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNPE01
Record Dates: First submitted 2023-12-19; First posted 2024-01-03 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Embolism; Acute Pulmonary Embolism; Cardiovascular Diseases; Venous Thromboembolism
Keywords: pulmonary embolism; aspiration thrombectomy; PE; catheter directed thrombectomy
MeSH Terms: conditions — Pulmonary Embolism; Cardiovascular Diseases; Venous Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Mechanical Thrombectomy via Cleaner Pro (Experimental): Participants will receive catheter-directed therapy via mechanical aspiration thrombectomy for the treatment of pulmonary embolism (PE) using the Cleaner Pro Thrombectomy System.
  Interventions: Device: Cleaner Pro Thrombectomy System

INTERVENTIONS:
Device: Cleaner Pro Thrombectomy System — The Cleaner™ Pro Thrombectomy System ("Cleaner Pro") is a catheter-based aspiration thrombectomy device comprised of a handpiece, an aspiration catheter, a dilator, and an aspiration canister.
  Other Names: Cleaner Vac Thrombectomy System

SUMMARY:
To evaluate the safety and efficacy of the Cleaner™ Pro Thrombectomy System for aspiration thrombectomy in patients with acute pulmonary embolism (PE).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at the time of consent
* Clinical signs, symptoms, and presentation consistent with acute PE
* Onset of PE symptoms occurred within 14 days of presentation
* Filling defect in at least one main or lobar pulmonary artery evidenced by CTA
* RV dysfunction on CTA or echocardiography defined as RV/LV ratio >0.9

Exclusion Criteria:

* tPA use within 14 days prior to baseline CTA
* Systolic BP <90 mmHg for 15 min or the requirement of inotropic support to maintain systolic BP ≥90 mmHg
* Diagnosis of pulmonary hypertension primary type I or CTEPH; if patient does not have diagnosis of pulmonary hypertension but peak PA >70 mmHg by right heart catheterization or elevated main pulmonary artery to aorta ratio (MPA:A), up to investigator discretion.
* History of severe or chronic pulmonary hypertension
* FiO2 requirement >40% or >6 LPM to keep oxygen saturations >90%
* Hematocrit <28%
* Platelets <100,000/µL
* Serum creatinine >1.8 mg/dL
* INR >3
* aPTT (or PTT) >50 seconds on no anticoagulation
* History of heparin-induced thrombocytopenia (HIT)
* Recent (within six months) history of stroke, transient ischemic attack (TIA), or intracranial bleeding
* Recent (within one month) history of active bleeding from a major organ
* Absolute contraindication to anticoagulation
* Major trauma such as head trauma, or other active intracranial, or intraspinal disease within 14 days
* Presence of intracardiac lead in the right ventricle or right atrium placed within 6 months
* Cardiovascular or pulmonary surgery within last 7 days
* Cancer which requires active chemotherapy
* Known serious, uncontrolled sensitivity to radiographic agents
* Life expectancy <90 days, as determined by investigator
* Female who is pregnant
* Intracardiac thrombus
* Patients who present with cardiac arrest and/or are on extracorporeal membrane oxygenation (ECMO) or ECMO required to perform interventional procedure
* Simultaneous participation in another investigational study
* Patients with known coagulation disorders such as antiphospholipid, Protein C, and Protein S
* Presentation of PE with paradoxical emboli which may be diagnosed by concurrent stroke or concurrent arterialization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2027-06-04 (Estimated); Study Completion 2027-09-02 (Estimated)

PRIMARY OUTCOMES:
Change in Right Ventricle (RV)/Left Ventricle (LV) Ratio | At 48 hours post-procedure
  Change in RV/LV ratio between baseline and 48 hours post procedure assessed by CTA.
Rate of Major Adverse Events (MAEs) | At 48 hours post-procedure
  Rate of MAEs within the first 48 hours after the index procedure, defined as:
  Device-related death Major bleeding, and Device-related Serious Adverse Events which includes clinical deterioration, pulmonary vascular injury, and cardiac injury.

SECONDARY OUTCOMES:
Rate of device-related complications and device-related death | Within 48 hours of the procedure
  Rate of device-related complications including major bleeding, clinical deterioration, pulmonary vascular injury, and cardiac injury, and device-related death within 48 hours of the index procedure.
Rate of device-related SAEs and all-cause mortality | Within 30 days of procedure
  Rate of device-related serious adverse events (SAEs) and death for any cause within 30 days post-procedure.
Rate of Symptomatic PE Recurrence | Within 30 days of the procedure
  Rate of Symptomatic PE recurrence within 30 days.
Volume of blood aspirated | At index procedure
  The amount of blood aspirated during the procedure.
Use of thrombolytics | Within 48 hours of the procedure
  Use of thrombolytics within 48 hours of the procedure.
Change in Modified Miller Index | At 48 hours post-procedure
  Change in Modified Miller Index between baseline and 48 hours post-procedure assessed by CTA. This index score quantifies arterial obstruction in pulmonary embolism. The higher the score, the more perfusion is reduced.
Quality of Life assessed via PEmb-QoL | At 30 days post-procedure
  Self-assessment of PE-related complaints and daily living limitations (including work and social). The PEmb-QoL measures 6 dimensions, with higher scores being worse.
Quality of Life assessed via EQ-5D-5L | At 30 days post-procedure
  Self-assessment of activities for daily living. The EQ-5D-5L measures 5 dimensions, with higher scores being worse.

CONTACTS AND LOCATIONS:
Overall Officials: Danyel C Carr, MS, Study Director — Argon Medical Devices; Pete J Stibbs, MD, Study Director — Argon Medical Devices
Locations (17):
- United States (17):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Medstar Health Research Institute, Washington D.C., District of Columbia
  - Ascension Sacred Heart Hospital, Pensacola, Florida
  - BayCare Health System, Tampa, Florida
  - Insight Hospital and Medical Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Ascension St. Vincent Hospital, Indianapolis, Indiana
  - UMass Chan Medical School, Worcester, Massachusetts
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - University at Buffalo, Buffalo, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Promedica Toledo Hospital, Toledo, Ohio
  - Ascension St. John Jane Phillips Medical Center, Bartlesville, Oklahoma
  - Ascension St. John Hospital, Tulsa, Oklahoma
  - Baylor Scott and White Heart and Vascular Hospital - Dallas, Dallas, Texas
  - Baylor Scott & White The Heart Hospital - Plano, Plano, Texas

IPD SHARING:
Plan to Share IPD: No